CLINICAL TRIAL: NCT01636856
Title: Effects of Oropharyngeal Exercises on Snoring Intensity, Symptoms, Upper Airway Anatomy and Collapsability of Upper Airway Awake and Asleep in Patients With Primary Snoring and Mild to Moderate Obstructive Sleep Apnea
Brief Title: Effects of Oropharyngeal Exercises on Patients With Primary Snore, Mild and Moderate Obstructive
Acronym: EOE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Geraldo Lorenzi-Filho, Associated Professor of Pulmonary Division, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3604/11/022
Record Dates: First submitted 2012-07-05; First posted 2012-07-10 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Primary Snore, Obstructive Sleep Apnea (Mild and Moderate).
Keywords: oropharyngeal exercises, obstructive sleep apnea, speech therapy, magnetic resonance, PCRIT, negative expiratory pressure, snore
MeSH Terms: conditions — Sleep Apnea, Obstructive; Lymphoma, Follicular; Communication Disorders; Snoring | interventions — Nasal Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Oropharyngeal exercises and oropharyngeal functions
  Interventions: Behavioral: Oropharyngeal exercises
- 2 (Sham Comparator): Nasal dilator, respiratory exercise, nasal lavage
  Interventions: Behavioral: Respiratory exercises, nasal dilator, nasal lavage

INTERVENTIONS:
Behavioral: Oropharyngeal exercises — Oropharyngeal exercises (derived from speech language pathology) to the soft palate, tongue and facial muscles exercises as well as stomatognathic functions.
  Arms: 1
Behavioral: Respiratory exercises, nasal dilator, nasal lavage — Respiratory exercises, nasal dilator, nasal lavage
  Arms: 2

SUMMARY:
Randomized study of patients with primary snore, mild and moderate obstructive sleep apnea. Protocol include 40 patients randomized to oropharyngeal exercise or use of nasal dilator, breathing exercise and nasal lavage. The objectives are study the effects of therapy on oropharyngeal in a series of clinical and physiologic and anatomic variables, changes on snore and quality of sleep using Pharyngeal Critical Pressure, Magnetic Resonance, Negative expiratory pressure and snore analyses. Hypothesis that the therapy group (oropharyngeal exercises) will have more modifications compared to the control group.

DETAILED DESCRIPTION:
This is randomized study with multiple primary endpoints. In December 2012 the study also started collecting tongue strength and endurance (IOPI). Because not all patients are able to perform all evaluations, the publications will be divided and presented according to the completion of the required number of patients for each primary endpoint.

ELIGIBILITY:
Inclusion Criteria:

subjects with primary snore, mild and moderate obstructive sleep apnea

Exclusion Criteria:

BMI > or = 40, craniofacial malformations, smokers, pregnant women, edentulous, total dental prostheses, use of hypnotic medications, stroke, neuromuscular dystrophy, coronary artery disease, chronic heart failure, chronic obstructive pulmonary disease, severe nasal obstructive disease, pharyngeal surgery,already made some kind of treatment for obstructive sleep apnea.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Upper airway collapsability | 3 months
Images from magnetic resonance | 3 months
Negative expiratory pressure | 3 months
Snore | 3 months

SECONDARY OUTCOMES:
Sleep related questionnaires | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Ieto, Principal Investigator — Heart Institute - InCor; Fabiane Kayamori, Principal Investigator — Heart Institute - InCor; Geraldo Lorenzi-Filho, MD, PhD, Principal Investigator — Heart Institute - InCor
Locations (1):
- Incor- Heart Institute, Sleep Laboratory, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Ieto V, Kayamori F, Montes MI, Hirata RP, Gregorio MG, Alencar AM, Drager LF, Genta PR, Lorenzi-Filho G. Effects of Oropharyngeal Exercises on Snoring: A Randomized Trial. Chest. 2015 Sep;148(3):683-691. doi: 10.1378/chest.14-2953. PMID 25950418